CLINICAL TRIAL: NCT02870283
Title: Assessment of Cost- Effectiveness Interventions and the Quality of Life in Patients With Mood Disorders Through Resources Available in Brazilian Public Health
Brief Title: Cost- Effectiveness and Quality of Life Assessment in Mood Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Flávia Barros da Silva Lima, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-013
Record Dates: First submitted 2016-05-26; First posted 2016-08-17 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2016-08

CONDITIONS: Bipolar Disorder
Keywords: Cost effectiveness; Bipolar disorder; Mixed episodes; Quality of life
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Valproic Acid; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lithium (Active Comparator): Subjects were randomized into three groups: (lithium, valproic acid, or carbamazepine).
  Group (A) Started Lithium (900mg-1500mg)
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  1. First step: Monotherapy with Lithium (900-1500mg) Non responsive patients: 2nd step.
  2. Second step: Randomization for lithium (900mg-1500mg) + valproic acid (1000mg-1500mg) OR lithium (900mg-1500mg) + carbamazepine (600mg-1200mg).
     Non responsive patients: 3rd step.
  3. Third step: Crossover lithium (900mg-1500mg) + valproic acid (1000mg-1500mg) X lithium (900mg-1500mg) + carbamazepine (600mg-1200mg).
     Non responsive patients: 4th step.
  4. Fourth step: Association with risperidone (1-6mg)
  Interventions: Drug: Lithium
- Acid Valproic (Active Comparator): Subjects were randomized into three groups: (lithium, valproic acid, or carbamazepine).
  Group (B) Started Valproic Acid (1000mg-1500mg).
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  1. First step: Monotherapy with Valproic Acid (1000mg-1500mg) Non responsive patients: 2nd step.
  2. Second step: Association with lithium (900mg-1500mg). Non responsive patients: 3rd step.
  3. Third step: Crossover: lithium (900mg-1500mg) + carbamazepine (600mg-1200mg). Non responsive patients: 4th step.
  4. Fourth step: Association with risperidone (1-6mg)
  Interventions: Drug: Valproic Acid
- Carbamazepine (Active Comparator): Subjects were randomized into three groups: (lithium, valproic acid, or carbamazepine).
  Group (C) Started Carbamazepine (600mg-1200mg).
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  1. First step: Monotherapy with Carbamazepine (600mg-1200mg). Non responsive patients: 2nd step.
  2. Second step: Association with lithium (900mg-1500mg). Non responsive patients: 3rd step.
  3. Third step: Crossover: lithium (900mg-1500mg) + valproic acid (1000mg-1500mg). Non responsive patients: 4th step.
  4. Fourth step: Association with risperidone (1-6mg)
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Lithium
  Other Names: carbolitium
  Arms: Lithium
Drug: Valproic Acid
  Other Names: depakene
  Arms: Acid Valproic
Drug: Carbamazepine
  Other Names: tegretol
  Arms: Carbamazepine

SUMMARY:
To evaluate the effectiveness of three systematic interventions for Bipolar Disorder (BD) mixed episodes using medications available in the Brazilian Public Healthcare System (SUS), and assessment of the quality of life of these patients.

A randomized pragmatic trial was conducted. An algorithm was developed for the treatment of episodes of bipolar mixed episodes.

DETAILED DESCRIPTION:
The study design was that of a pragmatic randomized clinical trial to evaluate the effectiveness of treatments for mood disorders in a public healthcare context in the city of Porto Alegre, in southern Brazil. The algorithm was originally developed for the treatment of mixed episodes by a Delphi panel of experts from psychiatric associations in Brazil. All subjects provided an informed consent form, in writing, in order to participate in the study protocol, which was approved by the institutional ethics committee.

Procedures and measurements of the study

The subjects under evaluation were selected and they followed the stages defined by the treatment protocol:

1. Sample selection by being referred from the primary healthcare clinics in the municipality;
2. Informative talk about mood disorders and the research, with the informed consent forms being provided to the subjects;
3. Screening for BD mixed episodes with the use of the Patient Health Questionnaire (PHQ-9), and Hypomanic Symptoms Checklist Brazilian Version (HCL -32-BV);
4. Diagnostic evaluation through the Mini International Neuropsychiatric Interview (MINI) and clinical interview for individuals with positive results in the screening instruments;
5. Baseline and demographic assessments using standardized semi-structured interviews in the first and second visits;
6. In each clinic visit, the severity of the symptoms were evealuated using the Clinical Global Impression Scale (CGI), Hamilton Rating Scale for Depression (HRSD), and Young Manic Rating Scale (YMRS);
7. Biweekly follow-up, changed to monthly after stabilization - with a maximum follow-up period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ages between 18 and 65;
2. BD current acute mixed episode;
3. total capacity to understand and respond to self-applied instruments;
4. the presence of symptoms in the last 30 days;
5. abstinence for at least 30 days for drug addicts.

Exclusion Criteria:

1. presence of Organic Brain Syndrome (OBS);
2. pregnancy or lactation;
3. criteria for psychiatric hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-05; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Fleck, PhD, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lima AF, Miguel SR, Cohen M, Zimmermann JJ, Shansis FM, Cruz LN, Ziegelmann PK, Polanczyk CA, Fleck MP. Effectiveness evaluation of mood disorder treatment algorithms in Brazilian public healthcare patients. Braz J Psychiatry. 2018 Jan-Mar;40(1):26-34. doi: 10.1590/1516-4446-2016-2147. Epub 2017 Aug 21. PMID 28832750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Response to treatment was assessed for the entire algorithm. There were no comparisons between the steps of each arm of the study
Groups:
- Lithium: Subjects were randomized into three groups: (lithium, valproic acid, or carbamazepine).
  Group (A) Started Lithium (900mg-1500mg)
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  1. First step: Monotherapy with Lithium (900-1500mg) Non responsive patients: 2nd step.
  2. Second step: Randomization for lithium (900mg-1500mg) + valproic acid (1000mg-1500mg) OR lithium (900mg-1500mg) + carbamazepine (600mg-1200mg).
     Non responsive patients: 3rd step.
  3. Third step: Crossover lithium (900mg-1500mg) + valproic acid (1000mg-1500mg) X lithium (900mg-1500mg) + carbamazepine (600mg-1200mg).
     Non responsive patients: 4th step.
  4. Fourth step: Association with risperidone (1-6mg)
  Lithium
- Acid Valproic: Subjects were randomized into three groups: (lithium, valproic acid, or carbamazepine).
  Group (B) Started Valproic Acid (1000mg-1500mg).
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  1. First step: Monotherapy with Valproic Acid (1000mg-1500mg) Non responsive patients: 2nd step.
  2. Second step: Association with lithium (900mg-1500mg). Non responsive patients: 3rd step.
  3. Third step: Crossover: lithium (900mg-1500mg) + carbamazepine (600mg-1200mg). Non responsive patients: 4th step.
  4. Fourth step: Association with risperidone (1-6mg)
  Valproic Acid
- Carbamazepine: Subjects were randomized into three groups: (lithium, valproic acid, or carbamazepine).
  Group (C) Started Carbamazepine (600mg-1200mg).
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  1. First step: Monotherapy with Carbamazepine (600mg-1200mg). Non responsive patients: 2nd step.
  2. Second step: Association with lithium (900mg-1500mg). Non responsive patients: 3rd step.
  3. Third step: Crossover: lithium (900mg-1500mg) + valproic acid (1000mg-1500mg). Non responsive patients: 4th step.
  4. Fourth step: Association with risperidone (1-6mg)
  Carbamazepine
Period: Overall Study
Arm/Group | Lithium | Acid Valproic | Carbamazepine
Started | 38 | 35 | 34
Completed | 35 | 26 | 15
Not Completed | 3 | 9 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium | Acid Valproic | Carbamazepine | Total
Number analyzed (Participants) | 38 | 35 | 34 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 34 | 107
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (13.17) | 43.6 (13.17) | 43.6 (13.17) | 43.6 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 27 | 86
  Male | 7 | 7 | 7 | 21
Region of Enrollment [Number; unit: participants]
  Brazil | 38 | 35 | 34 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Treatment"
Description: Response to treatment was defined as a 50% reduction from baseline scores in Hamilton Rating Scale for Depression (HRSD)and Young Mania Rating Scale (YMRS) scales HRSD was developed to evaluate and quantify depression.Its abbreviated version,. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal. The cutoff points are: 8-17 for mild depression,18-24 for moderate depression, and 25 or more for severe depression. The maximum score being 52 on the 17-point scale.
  YMRS is is the most widely used assessment tool for manic symptoms. The scale consists of 11 items .The YMRS follows the style of the Hamilton Rating Scale for Depression (HAM-D) with each item given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/agressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Scores of YMRS > 20 generates indicate mania
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium | Acid Valproic | Carbamazepine
Number analyzed (Participants) | 38 | 35 | 34
Participants | 31 | 28 | 27

2. Secondary Outcome: Number of Participants With Remission to Treatment
Description: The remission outcome was established as obtaining three consecutive visits with scores of values considered asymptomatic Hamilton Rating Scale for Depression(HRSD <7 points) and Young Mania Rating Scale (YMRS <6 points) during the trial. The subjects that were asymptomatic for at least 6-8 month were considered to be in partial remission and complete if at least 12 months without symptoms, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium | Acid Valproic | Carbamazepine
Number analyzed (Participants) | 38 | 35 | 34
Participants | 10 | 9 | 9

3. Secondary Outcome: Quality of Life - WHOQOL Bref Intrument
Description: Quality of Life - WHOQOL -BREF instrument scores scores 0-20 . higher scores mean a better outcome. The quality of life was assessed for entire algorithm. There were no comparisons between each arms of the study.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Acid Valproic | Carbamazepine
Number analyzed (Participants) | 35 | 26 | 15
score on a scale | 10.91 (3.44) | 10.91 (3.44) | 10.91 (3.44)

ADVERSE EVENTS:
Arm/Group | Lithium | Acid Valproic | Carbamazepine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/38 | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No